CLINICAL TRIAL: NCT00256022
Title: The Effect of Prophylactic Pre Operative Probiotic Therapy on Peri Operative Endotoxin Levels in Cardiac Surgery Patients.
Brief Title: The Effect of Prophylactic Pre Operative Probiotic Therapy on Endotoxin Levels in Cardiac Surgery Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to delays with logistics and protocol revision not viable to continue.
Sponsor: Melbourne Health (Other)
Collaborators: Intensive Care Unit Research Department, Royal Melbourne Hospital (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000.177
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-04

CONDITIONS: Preoperative Cardiac Surgery Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lactobacillus Acidophilus Arm (Active Comparator): The probiotic will be given to the patient 2 a dy for between 2-7 days preoperatively. Participation in this study requires 6 separate blood tests commencing at the start of surgery and continuing for 24 hours immediately post operatively.
  Interventions: Drug: Lactobacillus Probiotic
- Lactobacillus Fermentum Arm (Active Comparator): The probiotic will be given to the patient 2 a dy for between 2-7 days preoperatively. Participation in this study requires 6 separate blood tests commencing at the start of surgery and continuing for 24 hours immediately post operatively.
  Interventions: Drug: Lactobacillus Probiotic
- Lactobacillus Fermentum and Lactobacillus Acidophilus (Active Comparator): The probiotic will be given to the patient 2 a dy for between 2-7 days preoperatively. Participation in this study requires 6 separate blood tests commencing at the start of surgery and continuing for 24 hours immediately post operatively.
  Interventions: Drug: Lactobacillus Probiotic
- Placebo (Placebo Comparator): The placebo will be given to the patient 2 a day for between 2-7 days preoperatively. Participation in this study requires 6 separate blood tests commencing at the start of surgery and continuing for 24 hours immediately post operatively.
  Interventions: Other: Lactose Powder

INTERVENTIONS:
Drug: Lactobacillus Probiotic
  Arms: Lactobacillus Acidophilus Arm; Lactobacillus Fermentum Arm; Lactobacillus Fermentum and Lactobacillus Acidophilus
Other: Lactose Powder
  Arms: Placebo

SUMMARY:
The primary hypothesis for the study is that pre-operative prophylactic probiotic Lactobacilli tablets will reduce the severity and incidence of endotoxin rise in post cardiopulmonary bypass in cardiac surgery patients.

Endotoxins are large heat stable lipopolysaccharides, which are found in the cell wall of gram negative bacteria. It has been assumed that the intestinal bacteria are the primary source of the plasma endotoxin in cardiac surgery patients.Lactobacilli have been reported as effective in counteracting gram negative bacteria in the gut.Thus Lactobacilli may be effective in reducing the endotoxin rise associated with cardiopulmonary bypass, which may potentially reduce the incidence of the syndrome of generalised inflammation and low systemic vascular resistance post cardiopulmonary bypass.

DETAILED DESCRIPTION:
The study compare endotoxin levels of post operative cardiac surgery patients who have received pre operative prophylactic probiotic Lactobacillus tablets. Compared to patients who have received a placebo.

Two different lactobacillus strains will be assessed in the study: Lactobacillus Acidophilus and Lactobacillus Fermentum. There are 4 treatment groups in this study. Lactobacillus Acidophilus,Lactobacillus Fermentum, Lactobacillus Fermentum and Lactobacillus Acidophilus and Placebo.

The probiotic/placebo will be given to the patient 2 a dy for between 2-7 days preoperatively. Participation in this study requires 6 separate blood tests commencing at the start of surgery and continuing for 24 hours immediately post operatively.A total of 30 mls of blood is required.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cardiac surgery requiring cardiopulmonary bypass will be approached for consent to participate in the study.

Exclusion Criteria:

* Age greater than or equal to 18 years
* Current usage of a probiotic product
* Past history of asthma or recurrent urticaria, pregnancy, HIV infection, immunosuppression and pre existing intestinal disorder.

The Lactobacillus acidophilus preparation to be used in this study contains a very small amount of MSG (total dose 20mg/day, equivalent to 10% of the total dose used to test MSG sensitivity) and as a precaution patients with asthma or recurrent urticaria will be excluded. As the Lactobacillus preparation contains live micro organisms, immunosuppressed and pregnant patients will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variable of this study is endotoxin rise in the first 24 hours post commencement of surgery.

SECONDARY OUTCOMES:
The secondary outcomes include peak IL-6 levels, the development of post operative generalised inflammation and low systemic vascular resistance.

CONTACTS AND LOCATIONS:
Overall Officials: John F Cade, Principal Investigator — Intensive Care Unit, Royal Melbourne Hospital